CLINICAL TRIAL: NCT07146867
Title: Metabolic Responses to a Single Session of High-intensity Interval Training in Insufficiently Active Young Adults. Effects on Adiponectin Isoforms
Brief Title: Effects of One HIIT Session on Adiponectin Isoforms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Sebastián (Other)
Responsible Party: Principal Investigator, Sergio Martinez-Huenchullan, Researcher, Universidad San Sebastián
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AcuteHIIT
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Inactivity, Physical
Keywords: adiponectin; high intensity interval training
MeSH Terms: conditions — Sedentary Behavior | interventions — High-Intensity Interval Training; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High intensity interval training (Experimental): One session of high intensity interval training
  Interventions: Behavioral: High intensity interval training (exercise)

INTERVENTIONS:
Behavioral: High intensity interval training (exercise) — One 30 minute session of high intensity interval training

SUMMARY:
The goal of this observational quasi-experimental study is to evaluate whether a single session of high-intensity interval training (HIIT) can acutely modulate metabolic markers, particularly adiponectin isoforms, in insufficiently active young adults (men and women, 18-29 years, free of cardiometabolic disease).

The main questions it aims to answer are:

Does a single HIIT session increase circulating medium- and high-molecular-weight adiponectin?

Does HIIT acutely alter lipid and glucose metabolism markers such as non-HDL cholesterol, insulin, and lactate?

Participants completed the following tasks:

Underwent baseline assessments (anthropometry, body composition, and resting cardiovascular parameters).

Performed one HIIT session consisting of six 3-minute intervals at 80% heart rate reserve, each followed by 3 minutes of active recovery.

Provided blood samples before and immediately after exercise to analyze adiponectin isoforms (LMW, MMW, HMW) via Western blot and to measure glucose, insulin, lipid profile, liver enzymes, and lactate.

Summary of findings:

A single HIIT session significantly increased medium-molecular-weight adiponectin (~19%), decreased the HMW/MMW ratio, and elevated lactate and non-HDL cholesterol. No significant changes were observed in LMW or HMW adiponectin. These results suggest that MMW adiponectin is an early, sensitive marker of acute exercise response in sedentary young adults, though further research is needed to confirm long-term implications

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 29 years, engage in less than 150 minutes of moderate-intensity or 75 minutes of vigorous-intensity physical activity per week), and having no positive responses on the PAR-Q & YOU questionnaire

Exclusion Criteria:

* diagnosis of cardiometabolic disease or the use of anti-inflammatory treatment during the week prior to participation

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Adiponectin isoforms | Before and immediately after the exercise session
Adiponectin isoforms | Before and immediately after the exercise session (30 minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad San Sebastián, Valdivia, Los Ríos Region, Chile

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Derived] Alvarado-Carrasco D, Gonzalez-Maraboli A, Reyes-Montalva M, Videla-Aguilar J, Bentes A, Penailillo L, Sandoval V, Martinez-Huenchullan S. Acute effects of high-intensity interval training on adiponectin isoforms in inactive young adults: a quasi-experimental study. BMC Sports Sci Med Rehabil. 2025 Dec 30;17(1):387. doi: 10.1186/s13102-025-01433-7. PMID 41469733

DOCUMENTS (1):
  • Informed Consent Form (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT07146867/ICF_000.pdf